CLINICAL TRIAL: NCT05480891
Title: Repurposing Transnasal Esophagoscopy: Targeting Interventions for a Community That Has Been Targeted for Cancer Risk
Brief Title: Transnasal Esophagoscopy (TNE) Esophageal Cancer Screening
Status: Terminated | Type: Observational
Why Stopped: Transnasal Esophagoscopy (TNE) scope is no longer manufactured so the study is unable to be continued.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Principal Investigator, H Steven Sims, Francis L. Lederer Professor, Otolaryngology - Head and Neck Surgery Director, The Chicago Institute for Voice Care (CIVC), University of Illinois at Chicago
Other Study IDs: 2022-0115
Record Dates: First submitted 2022-07-20; First posted 2022-07-29 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Transnasal Esophagoscopy (TNE) — While seated in an upright position a topical numbing medicine will be sprayed in your nose and the back of your throat.
  A thin, flexible tube less than ¼ inch in diameter, will be placed in one of your nostrils and advanced to the back of your throat. When the tube reaches the back of the throat you will be asked to drink sips of water to help move the tube into and down the esophagus as it is advanced. The tip of the tube has a small light and camera built in that allows the doctor to see the structures of the mouth and esophagus as the tube is advanced. Once the tube is in the esophagus, the physician will examine your esophagus for any abnormal changes.
  Once the visual inspection is complete the tube will be gently removed through your nose. The procedure will take approximately 10-15 minutes of time.

SUMMARY:
This research study is being done for 2 reasons: 1) The investigators want to learn about the eating, smoking and drinking habits of adults, 18 years of age and older, in various Chicago communities, and 2) the investigators want to offer screening for participants whose smoking and drinking habits put them at risk for cancer.

DETAILED DESCRIPTION:
There are longstanding disparities in healthcare outcomes in the United States. These differences often correlate from the effects of structural racism and how this factor has shaped healthcare in our society.

Esophageal cancer presents as one of two distinct histological cell types, adenocarcinoma and squamous cell carcinoma (SCC). The majority of White patients presenting with esophageal cancer are diagnosed with adenocarcinoma while Black and non-caucasian patients are more commonly diagnosed with squamous cell carcinoma. The detection and treatment of these two types of esophageal cancers vary.

Trans-nasal esophagoscopy (TNE) is used primarily to assess chronic acid reflux as well as Barrett's esophagus, both symptoms being associated with adenocarcinoma. The use of TNE for disease screening offers the opportunity for early diagnosis and treatment of esophageal adenocarcinoma. Currently there is no parallel method of screening and diagnosis for patients with the potential for squamous cell carcinoma (SCC).

In an effort to decrease the disease identification, diagnosis, and treatment gap between these populations, this study will evaluate the use of TNE as a screening tool for African-Americans and non-caucasian patients with high risk factors associated with the development of esophageal SCC.

All adult patients 18 years of age and older will be asked to participate in a survey at one of the UI Health community health centers. The survey will include questions about smoking and alcohol consumption habits, which have been shown to be specific risk factors associated with esophageal SCC. Additional information, such as the use of mentholated cigarettes and fortified wines will be surveyed as such products are selectively marketed in African American communities and may increase the prevalence of SCC in these communities. Following review of the survey results from the health centers, all patients presenting with a dysphasia or difficulty swallowing, and patients who are 40 years of age and older and who have been determined to be high risk for SCC based on their survey results, will be offered the opportunity to have a TNE screening for esophageal cancer. Data gathered as a result of the study will be shared with participating communities and with medical health providers in an effort to improve patient knowledge and access to quality healthcare.

There are longstanding, historical, and current disparities in healthcare outcomes in the United States.[1-4] While we often classify these differences as racial, they are more likely to correlate with the effects of systemic racism that manifest as societal determinants of health. Segregation, whether legally sanctioned or de facto, molds the composition of neighborhoods and significantly influences access to quality healthcare.

Esophageal cancer incidence, stage at diagnosis, and mortality is one disease process that highlights these discrepancies. This year, an estimated 19,260 adults, most of whom are expected to be males, will be diagnosed with esophageal cancer. The two major types of esophageal cancer are adenocarcinoma and squamous cell carcinoma. In the United States, esophageal cancer is more common in Caucasians than African Americans/non-Caucasians. In Caucasians the disease is frequently diagnosed as an adenocarcinoma, which implies the cancer arose from gland producing cells in the body. Squamous cell carcinoma, which originates from skin cells and mucosal linings in the body, is more common in the African American/non-Caucasian populations.

The five-year survival rate for esophageal cancer was reported to be five per cent four decades ago. Today the survival rate has improved to approximately twenty per cent. However, in 1970, the survival rate for White males was approximately four times that of Black/non-caucasian males, and in 2021, that ratio persists. Simply stated, Black and non-caucasian men are more likely to die from squamous cell cancer (SCCA) of the esophagus than any other demographic in the United States. The reason for the disparity in survival rates may be the result of a more proactive early screening process in the White population as symptoms arise. Adenocarcinoma, the more common form of esophageal cancer in the Caucasian population is frequently associated with Gastro-Esophageal Reflux Disease (GERD) or Barrett's esophagus. Early screenings and diagnosis of these two precursor causes of adenocarcinoma allows for early detection and treatment, thereby decreasing mortality. [8,9,19] Survival of esophageal cancer is associated with disease stage at diagnosis. Five-year survival is nearly 50% if the disease is diagnosed early and has not metastasized to lymph nodes or surrounding tissues or organs. Once the cancer has spread to lymph nodes, the average rate of survival is approximately 25%. If the cancer is not diagnosed until it has spread to other, more distant parts of the body, survival is estimated to be around 5%.

Trans-nasal esophagoscopy (TNE) is currently used primarily to assess chronic acid reflux as well as to screen for Barrett's esophagus. Clinicians have tended to employ this screening tool to look for changes that could lead to adenocarcinoma of the esophagus in response to symptoms. Caucasian males over age 50 are the primary target group for the current screening paradigm. Published reports and guidelines for the use of TNE as a screening tool for adenocarcinoma are readily available to the medical community. Patients, once diagnosed for GERD or Barrett's esophagus have annual visits with a gastroenterologist for sustained screening. Conversely, African-American/non-caucasian males who are considered at lower risk for Barrett's esophagus may not be referred for screening surveillance. The fact that African-American and non-caucasian males, particularly those with a history of alcohol and tobacco consumption, may be at increased risk for esophageal squamous cell carcinoma has not led to a specific screening protocol for this patient population. In fact, certain risks, such as mentholated cigarettes and fortified wines, which are selectively marketed in non-caucasian communities, may be a major factor in the increased prevalence and severity of SCC in these specific communities.

This study aims to evaluate the use of TNE as a screening tool for targeted populations with known risk factors for esophageal SCC. Specific symptoms are considered for the use of TNE for the diagnosis and treatment of esophageal adenocarcinoma, which is most prevalent in white males. This study aims to evaluate a more extensive use of TNE as a screening tool for at risk African American/non-Caucasian populations for the early diagnosis and treatment of esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age or older
* Patients being seen at one of the UI Health Centers for an ear, nose, or throat related concern.
* Patients who have a history of both smoking and drinking.
* Patients must be willing to complete a study survey.
* Patients must understand the purpose and procedures of the study and be willing to participate.
* Patients who speak English.
* All adult men and women who meet the study criteria will be asked to participate in the study without regard to race, gender or socioeconomic status.
* For Part 2 of the study, inclusion criteria includes all patients 40 and over with a history or smoking and drinking as well as patients 18 years of age and older who present with dysphasia and/or pain when swallowing. Patients eligible for Part 2 of the study will be informed of the study, but they will not be consented during their clinic visit.

Exclusion Criteria:

* Male and Female patients under the age of 18.
* Patients who are not being seen at one of the UI Health Community Health
* Centers for an ear, nose or throat related concern.
* Patients who do not have a history of both drinking and smoking.
* Patients unwilling to complete the study survey.
* Women who are pregnant will be excluded from both Part 1 and Part 2 of the study.
* Patients unable to understand the purpose and procedures of the study and/or who are not willing to participate.
* Patients who do not speak English.

Excluded or Vulnerable Populations

* Minors will be excluded from the study because they are not at risk for the factors being studied in the research.
* Subjects who are not English speaking will be excluded due to the limited capacity of the primary investigators to obtain informed consent in this population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be recruited from UI Health Mile Square Community Health Centers, a Federally Qualified Health Center (FQHC). Mile Square has always been committed to serving Chicago's disenfranchised communities. Patients are predominantly minority; many of whom are at or below the Federal Poverty Level and have public insurance or are uninsured. The Mile Square system provides comprehensive primary care for children and adults. The system includes primary care clinics, as well school-based health centers and nurse-practice sites that provide health care for people with severe and persistent mental illness.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Conduct a population survey of UI Health and Mile Square Community Center patients focusing on specific risk factors associated with esophageal squamous cell carcinoma (ESCC) | Through study completion, an average of 2 years
  The researchers will collect data on the consumption of alcohol and tobacco as they are known risk factors for ESCC. The researchers will specifically assess consumption of fortified wines and mentholated cigarettes based on the targeted marketing of these products in identified communities. The researchers will also assess consumption of fresh fruits and vegetables and proportion of fat in dietary consumption to assess whether these conditions are associated with cancer risk.
Develop risk/screening criteria for esophageal squamous cell carcinoma in at risk populations | Through study completion, anticipating 2 years
  The researchers hope our data will serve to help create a risk stratification that can parallel current guidelines for screening patients for adenocarcinoma (which primarily affects Caucasian males). The researchers will compare results of trans-nasal esophagoscopy (TNE) exam and any biopsy specimens collected with the risk profile generated by survey results.
community education | Ongoing throughout the study, approximately 2 years
  The design of this study includes partnership with the at-risk community to engage in education about the stated risk factors and promote preventive health and encourage participation in screenings.

CONTACTS AND LOCATIONS:
Overall Officials: H. Steven Sims, MD, Principal Investigator — University of Illinois Chicago
Locations (2):
- United States (2):
  - Mile Square Health Center-University of Illinois Hospital, Chicago, Illinois
  - University of Illinois, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No